CLINICAL TRIAL: NCT04192123
Title: A Prospective, Monocentric, Open-Label Test of the HM242 Wound and Irrigation Solution and Gel on Healthy Skin to Evaluate Safety and Local Tolerability
Brief Title: Open-Label Test of the HM242 Medical Devices to Evaluate Safety and Local Tolerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPM-G-H-1902
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Intact Skin
Keywords: Physical rinsing; Cleansing solution; Wound bed preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All patients will receive an occlusive patch per test treatment as follows:
  * Treatment 1: HM242-Solution
  * Treatment 2: HM242-Gel
  * Treatment 3: HM242-Solution and HM242-Gel
  * Treatment 4: Irritant control (sodium lauryl sulfate (SLS))
  * Treatment 5: Negative control
  Interventions: Device: HM242

INTERVENTIONS:
Device: HM242 — HM242-Solution and HM242-Gel will be topically applied in an occlusive patch for 48h on healthy skin on the subject's outer part of the upper arm.

SUMMARY:
It is the first clinical study aimed at assessing the safety and tolerability of HM242-Solution and HM242-Gel after their application under occlusion on intact skin. The HM242-Solution is intended for chronic wounds (e.g. pressure, venous leg and diabetic foot ulcers). The HM242-Solution should be used for physical rinsing and cleansing and subsequent decolonization of the wound prior to treatment with hydrogels and dressings. The HM242-Gel is a hydrogel for wound bed preparation to support the healing of the skin due to cleansing, moistening and subsequent decolonization and the coating of the wound.

The study will be conducted in outpatient manner, adult patients who are healthy and has an intact skin.

This is an prospective, open label, monocentric study. No comparative control group is planned as no other preventing infection solution is commercially available at this time.

DETAILED DESCRIPTION:
The objective of this study is to assess the local tolerability and safety of HM242-Solution and HM242-Gel after their application under occlusion on intact skin.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male or female subjects aged ≥ 18 years and ≤ 65 years.
* Healthy skin on the upper arms
* Skin type visually assessed from pale white to light brown
* Females with childbearing potential must have a negative urine pregnancy test at baseline and must agree to use a highly effective method of contraception for the duration of the clinical investigation.
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial prior to any trial-related activity and that all information has been understood

Exclusion Criteria:

* Breastfeeding or pregnant women
* Extremely tanned skin that may interfere with the tolerability assessment based on Investigator judgment
* Subjects with known or suspected allergies or skin hypersensitivity (e.g. acute dermatitis)
* Subjects with known or suspected allergies or hypersensitivity to any of the components of the Investigational Medical Devices
* Any illness or circumstance that could affect the trial purpose in the opinion of the investigator (e.g. intensive UV exposure)
* Dermatologic diseases or skin conditions (e.g. tattoos, multiple birth marks in the test area) that might interfere with the evaluation of test site reaction
* Within 3 weeks prior to Day 1 and during the entire trial: Any systemic or topical medication or therapy likely to interfere with the trial purposes: e.g. immune-modulating or immunosuppressive therapy (e.g. corticosteroids, cytotoxics, cyclosporine or radiotherapy).
* Within 7 days prior to Day 1 and during the entire trial: any topical dermatological agents applied on the upper arms (drugs or medical device), except usual skin care preparations and skin cleansing preparations like anionic tensides, cleansing soaps ointments, oils, enzymes, etc. (not allowed on test areas during the trial)
* During the entire trial: exposure to sunlight that could lead to sunburns or photo sensibilization reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of related Adverse Events from Study Start until the End of Study (EoS) | Day 1 to Day 10
  to assess safety of HM242-Solution and HM242-Gel in healthy subjects which will be assessed in terms of related adverse events occurrence during the study (as reported by subjects and/or observed by the investigator)

SECONDARY OUTCOMES:
Post treatment assessment (via patch test scoring system provided by International Contact Dermatitis Research Group) by the Investigator. Scoring system: "-" no reaction; "Ir" irritative reaction (vesicles, blister, necrosis) | Day 3, Day 4, Day 5
  to assess local tolerability of HM242-Solution and HM242-Gel in healthy subjects which will be assessed by the investigator using the patch test

CONTACTS AND LOCATIONS:
Overall Officials: Welf Prager, Dr. med, Principal Investigator — Dermatologische Praxis Prager & Partner
Locations (1):
- Dermatologische Praxis Prager & Partner, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No